CLINICAL TRIAL: NCT02823717
Title: Obstetric and Proctology Support of Patients With Perineums Suits. Prospective Cohort
Brief Title: Obstetric and Proctology Support of Patients With Perineums Suits
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: PERINEE COMPLET
Record Dates: First submitted 2016-06-29; First posted 2016-07-06 (Estimated); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Obstetric Complications; Muscle Tear

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Perineal tear grade III and IV are relatively common (1-10% of deliveries depending on the series), and are a source of potentially serious complications, even long time after delivery (especially disorders of anal continence, psychological trauma). If a number of risk factors are well described, the support arrangements at the time of delivery and the characteristics of the review Proctological remote delivery and its relationship to the clinical status of patients is little known and rarely studied.

In maternity wards of the hospital Saint Joseph Paris and Cochin-Port Royal group, patients with a diagnosis of severe perineal tear was made are taken following load with common rules, both for the immediate repair for the remote monitoring. Patients of both sites are indeed encouraged to consult in proctology consultation in Saint Joseph 4-6 months of birth.

The same support on both sites allows to consider the creation of a relatively homogeneous cohort in terms of support and consider an important recruitment. Moreover, the geographical proximity of the inclusions sites (maternity) with proctology service is likely to limit the risk of lost sight of.

DETAILED DESCRIPTION:
Main objective / secondary:

Describe exactly the operational management of severe perineal tear (grade III and IV), their context and the factors associated with them occurring, the results of clinical and paraclinical proctology examination carried away from the birth, and study their relationship with the clinical status of patients at 6 months, 1, 2 and 3 years of confinement.

Methodology :

Type prospective, multicentre, non-interventional Study duration: 6 years

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 years
* Affiliated to the national system of social security,
* Giving birth during the period of inclusion of the St. Joseph site or Port Royal for whom the diagnosis of severe perineal tear was done.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In maternity wards of the hospital Saint Joseph Paris and Cochin-Port Royal group, patients with a diagnosis of severe perineal tear was made are taken following load with common rules, both for the immediate repair for the remote monitoring. Patients of both sites are indeed encouraged to consult in proctology consultation in Saint Joseph 4-6 months of birth.
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2015-01-31 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of change of Bristol Score | 6 months, 1, 2 and 3 years of birth
  The Bristol stool scale is a diagnostic medical tool designed to classify the form of human faeces into seven categories. It is used in both clinical and experimental fields.
Assessment of change of anal incontinence score | 6 months, 1, 2 and 3 years of birth
  The severity of fecal incontinence can be assessed by a scoring system which takes into account the type and frequency of incontinence as well as the extent to which it alters the patient's life. This can also be used to monitor the patient over time, especially after interventions.

CONTACTS AND LOCATIONS:
Overall Officials: AZRIA Elie, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Ile-de-Francfe, France